CLINICAL TRIAL: NCT04288323
Title: Abbreviated MRI (AMRI) vs. Ultrasound for HCC Surveillance in Cirrhosis
Brief Title: Gadolinium Contrast-enhanced Abbreviated MRI (AMRI) vs. Standard Ultrasound for Hepatocellular Carcinoma (HCC) Surveillance in Patients With Cirrhosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Claude Sirlin, Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 171769
Record Dates: First submitted 2020-02-25; First posted 2020-02-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Liver Cancer; Liver Cirrhoses; Liver Carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — gadolinium ethoxybenzyl DTPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Experimental): This is a single arm study in which all participants have one ultrasound and one abbreviated MR exam
  Interventions: Drug: Gadolinium ethoxybenzyl diethylenetriamine pentaacetic acid

INTERVENTIONS:
Drug: Gadolinium ethoxybenzyl diethylenetriamine pentaacetic acid — This study involves an on-label use of Gadolinium ethoxybenzyl diethylenetriamine pentaacetic acid for the ....

SUMMARY:
This study compares gadolinium contrast-enhanced Abbreviated MRI (AMRI) to standard ultrasound for Hepatocellular Carcinoma (HCC) screening and surveillance in subjects with liver cirrhosis.

DETAILED DESCRIPTION:
Ultrasound (US) is currently used for HCC surveillance. However, US has certain limitations, so physicians use contrast CT or MRI. However, these are expensive and time-consuming procedures. We introduced an abbreviated MRI (AMRI) exam, which works well in cirrhotic and obese patients (unlike US), involves no ionizing radiation (unlike CT), and is rapid (unlike multi-phasic MRI) with total scanner times of less than ten minutes, and can be performed at about the same cost as US. This study in adult patients with cirrhosis will compare the performance of AMRI vs. US for detection of early-stage disease, and will help to define and validate a novel, rapid, accurate, and potentially cost-effective imaging protocol for HCC screening in high-risk individuals.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been fully informed and has personally signed and dated the written Informed Consent and Health Insurance Portability and Accountability Act (HIPAA) documents.
* Adult subjects of any gender and any ethnic group with liver cirrhosis of any etiology,
* Subject is able and willing to complete required research procedures (screening/enrollment, clinical evaluation, safety procedures, lab collection if needed, research AMRI exam, research US exam) and the three optional surveys (if subject opts in for that) within specified time windows, and is willing to allow the study team to review clinical data including but not limited to other clinical radiology reports and images.

Exclusion Criteria:

* VA patient
* < 18 years of age
* History of any liver cancer
* MRI contraindication(s)
* Subject knows that she is pregnant or states she trying to become pregnant
* Positive urine pregnancy test in woman of childbearing potential
* Nursing mother
* Subject has known allergy to any gadolinium agent
* Does not meet UC San Diego Intravenous Contrast Media Guidelines for administration of Eovist*
* Clinical screening exam of the liver performed at UCSD within the prior 90 days to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2025-12-16 (Actual)

PRIMARY OUTCOMES:
Comparison of full AMRI, simulated unenhanced AMRI, and US for HCC detection | up to one year
  per-patient sensitivity, specificity, positive predictive (PPV), negative predictive value (NPV) and accuracy of full AMRI vs. simulated unenhanced AMRI vs. US for HCC screening
Reader reliability of screening modalities | up to 12 months from completion of imaging
  the inter- and intra-reader reliability of full AMRI vs. simulated unenhanced AMRI vs. US for HCC screening

CONTACTS AND LOCATIONS:
Overall Officials: Claude B Sirlin, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No